CLINICAL TRIAL: NCT03114605
Title: imPact Of a mindfuLness-based Intervention on Quality of Life and reduCtion of Burnout Symptoms in policE Officers - the POLICE Study
Brief Title: Mindfulness-based Intervention in Police Officers - the POLICE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Centro Mente Aberta de Mindfulness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60406416.9.1001.5327; 160491 (Other: HCPA)
Record Dates: First submitted 2017-03-21; First posted 2017-04-14 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2017-03

CONDITIONS: Mindfulness; Police; Quality of Life; Burnout Syndrome
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Mindfulness-based Intervention (8 sessions - 2 hours each- 1 session/week)
  Interventions: Behavioral: Mindfulness-based Intervention
- Control (No Intervention): Waiting List

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention
  Arms: Mindfulness

SUMMARY:
The physical, emotional, economic and social damage of stress in the police corporation indicates an urgent call for preventive programs to approach stress reduction, burnout symptoms and promotion of quality of life and well-being.

The aim of the POLICE study is to evaluate the effectiveness of a Mindfulness-based intervention (MBI), compare to a waiting list (WL), in promoting quality of life and mental health in police officers.

DETAILED DESCRIPTION:
Police officers are submitted to a high burden of chronic stress. It is no surprise to find that this occupation ranks highest on diseases and accidents rates among all professions. These professionals presents a very high incidence of depression, anxiety disorders, alcohol dependence and suicidal behavior. In addition to mental health suffering, evidence suggests an increase risk of sudden cardiac death, diabetes, obesity and metabolic syndrome.

Mindfulness-based interventions have been tested and incorporated for several clinical and non-clinical conditions for more than three decades, with emphasis on stress reduction, promotion of quality of life, chronic pain, anxiety, depression and eating disorders.

The main hypothesis is that mindfulness training will improve their quality of life and reduce burnout symptoms. The investigators expect that individuals allocated in the MBI group will report, besides showing a better quality of life, mental health and less burnout, lower levels of stress, anxiety and depression symptoms.

With regard to the working mechanism of the MBI, investigators will examine if the changes in mindfulness trait, self-compassion, spirituality, decentering and resilience skills will mediate the main hypothesis.

The study will be conducted in Porto Alegre-RS and São Paulo-SP.

ELIGIBILITY:
Inclusion Criteria:

* Active Police Officers
* Availability to attend 8 sessions
* Willingness to voluntarily participation

Exclusion Criteria:

* Manic or hypomanic episode (current)
* Psychotic syndrome (current or past)
* Substance Use Disorder (past 12 months, except tobacco)
* Risk of suicide
* Previously completed Mindfulness-Based Intervention

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of Life | 8 weeks and 6 months
  A mindfulness intervention increase quality of life (measured by change in Whoqol-Bref scale).
Change from baseline burnout symptoms | 8 weeks and 6 months
  A mindfulness intervention decrease burnout symptoms (measured by change in MBI-GS scale)

SECONDARY OUTCOMES:
Change from baseline stress levels | 8 weeks and 6 months
  A mindfulness intervention decreases stress levels (measured by change in PSQ scale)
Change from baseline anxiety and depression symptoms | 8 weeks and 6 months
  A mindfulness intervention reduces anxiety and depression symptoms (measured by change in HADS scale)
Change from baseline Mental health | 8 weeks and 6 months
  A mindfulness intervention increases mental health (measured by change in GHQ-12 scale)
Change from baseline decentering skills | 8 weeks and 6 months
  A mindfulness intervention increases decentering skills (measured by change in EQ scale)
Change from baseline resilience | 8 weeks and 6 months
  A mindfulness intervention increases resilience capacity (measured by change in CD-RISC-25 scale)
Change from baseline spirituality, religiosity, personal beliefs | 8 weeks and 6 months
  A mindfulness intervention increases spirituality, religiosity and personal beliefs (measured by change in WHOQOL-SRPB-BREF scale)
Change from baseline religiosity | 8 weeks and 6 months
  A mindfulness intervention increases religiosity (measured by change in DUREL scale)
Change from baseline mindfulness trait | 8 weeks and 6 months
  A mindfulness intervention increases mindfulness trait (measured by change in MAAS scale)
Change from baseline self-compassion | 8 weeks and 6 months
  A mindfulness intervention increases self-compassion (measured by change in SCS scale)
Change from baseline Burnout subtypes | 8 weeks and 6 months
  A mindfulness intervention decrease burnout symptoms according to burnout subtypes (measured by change in BCSQ-12 scale)
Mindfulness mechanisms | 6 months
  Self-compassion (SCS scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers
Mindfulness mechanisms | 6 months
  Resilience capacity (CD-RISC-25 scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers
Mindfulness mechanisms | 6 months
  Decentering skills (EQ scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers
Mindfulness mechanisms | 6 months
  Spirituality (WHOQOL-SRPB-BREF scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers
Mindfulness mechanisms | 6 months
  Religiosity (DUREL scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers
Mindfulness mechanisms | 6 months
  Mindfulness trait (MAAS scale) will mediate quality of life enhancement and burnout symptoms reduction in police officers

CONTACTS AND LOCATIONS:
Overall Officials: Neusa Sica da Rocha, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Marcelo Marcos Piva Demarzo, MD, PhD, Principal Investigator — UNIFESP - Federal University of Sao Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trombka M, Demarzo M, Campos D, Antonio SB, Cicuto K, Walcher AL, Garcia-Campayo J, Schuman-Olivier Z, Rocha NS. Mindfulness Training Improves Quality of Life and Reduces Depression and Anxiety Symptoms Among Police Officers: Results From the POLICE Study-A Multicenter Randomized Controlled Trial. Front Psychiatry. 2021 Feb 26;12:624876. doi: 10.3389/fpsyt.2021.624876. eCollection 2021. PMID 33716824
- [Derived] Trombka M, Demarzo M, Bacas DC, Antonio SB, Cicuto K, Salvo V, Claudino FCA, Ribeiro L, Christopher M, Garcia-Campayo J, Rocha NS. Study protocol of a multicenter randomized controlled trial of mindfulness training to reduce burnout and promote quality of life in police officers: the POLICE study. BMC Psychiatry. 2018 May 25;18(1):151. doi: 10.1186/s12888-018-1726-7. PMID 29801444